CLINICAL TRIAL: NCT02680691
Title: The Effect of Robot Assisted Gait Training in Patients With Infratentorial Stroke
Brief Title: Robot Assisted Gait Training in Patients With Infratentorial Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Rehabilitation Center, Seoul, Korea (Other Government)
Responsible Party: Principal Investigator, Joon-Ho Shin, Team manager, National Rehabilitation Center, Seoul, Korea
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NRC-2015-01-002
Record Dates: First submitted 2016-02-09; First posted 2016-02-11 (Estimated); Last update posted 2018-03-05 (Actual); Status verified 2018-03

CONDITIONS: Stroke
Keywords: infratentorial stroke; robot; postural balance; Rehabilitation
MeSH Terms: conditions — Stroke | interventions — Congresses as Topic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Robot, then conventional training (Experimental): Robot assisted gait training 4 weeks after conventional gait training
  Interventions: Other: Robot, then conventional training
- Conventional, then robot training (Active Comparator): Conventional gait training 4 weeks after robot assisted gait training
  Interventions: Other: Conventional, then robot training

INTERVENTIONS:
Other: Robot, then conventional training — Robot assisted gait training from the baseline, then conventional gait training at 4 weeks after baseline
  Arms: Robot, then conventional training
Other: Conventional, then robot training — Conventional gait training from the baseline, then robot assisted gait training at 4 weeks after baseline
  Arms: Conventional, then robot training

SUMMARY:
The Effect of Robot Assisted Gait Training in Patients With Infratentorial Stroke

DETAILED DESCRIPTION:
The hypothesis is to determine the robotic gait training would be better than conventional therapy regarding the postural balance.

ELIGIBILITY:
Inclusion Criteria:

* Patients with infratentorial stroke
* Cognitively intact enough to understand and follow the instructions from the investigator

Exclusion Criteria:

* chronic neurological pathology
* orthopedic injuries
* femur lengths of less than 34cm
* severely limited range of lower extremity joint motion
* medical instability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2015-04; Primary Completion 2016-03 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Berg Balance Scale at 4 Weeks | Baseline and 4 weeks from baseline
  Berg Balance Scale assess the functional balance ability of participants with observation of 14 tasks, representing functional movements common in daily life

SECONDARY OUTCOMES:
Berg Balance Scale | Baseline, 4 weeks from baseline, 8 weeks from baseline, 12 weeks from baseline
  Berg Balance Scale assess the functional balance ability of participants with observation of 14 tasks, representing functional movements common in daily life
Trunk impairment scale | Baseline, 4 weeks from baseline, 8 weeks from baseline, 12 weeks from baseline
  Trunk impairment scale performs to evaluate the sitting balance and trunk control ability examining static sitting balance, dynamic sitting balance, and coordination
Functional Ambulation Category | Baseline, 4 weeks from baseline, 8 weeks from baseline, 12 weeks from baseline
  Categorizes patients according to basic motor skills necessary for functional ambulation. It represents the status of ambulation
10m walk test | Baseline, 4 weeks from baseline, 8 weeks from baseline, 12 weeks from baseline
  10m walk test is used to examine gait speed, in which participant was asked to walk on a 14 meter of walkway wearing harness with two conditions; with the fastest speed or with self-selected comfortable speed
Fugl-Meyer Assessment | Baseline, 4 weeks from baseline, 8 weeks from baseline, 12 weeks from baseline
  Fugl-Meyer Assessment uses to examine the motor function and coordination of affected lower extremity
Korean version of Falls efficacy scale | Baseline, 4 weeks from baseline, 8 weeks from baseline, 12 weeks from baseline
  Asseses perception of balance and stability during activities of daily living Assesses fear of falling in the elderly population
Scale for the assessment and rating of ataxia | Baseline, 4 weeks from baseline, 8 weeks from baseline, 12 weeks from baseline
  Scale for the assessment and rating for infratentorial stroke
Balance test using force plate | Baseline, 4 weeks from baseline, 8 weeks from baseline, 12 weeks from baseline
  Each subject performs the following four tasks resembling Romberg test: standing with their feet positioning with the distance between their shoulders with eyes open (FSEO) or closed (FSEC), and standing with their feet together with eyes open (FTEO) or closed (FTEC). Each task is performed for 20 seconds and repeat for three times.

CONTACTS AND LOCATIONS:
Overall Officials: Joon-Ho Shin, MS, Principal Investigator — National Rehabilitation Center
Locations (1):
- National Rehabilitation Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim HY, Shin JH, Yang SP, Shin MA, Lee SH. Robot-assisted gait training for balance and lower extremity function in patients with infratentorial stroke: a single-blinded randomized controlled trial. J Neuroeng Rehabil. 2019 Jul 29;16(1):99. doi: 10.1186/s12984-019-0553-5. PMID 31358017
- See also: Site of the present study — http://nrc.go.kr